CLINICAL TRIAL: NCT03893266
Title: Exploratory Study of the Needs of Type 1 Diabetic Patients in Therapeutic Education in Order to Reconcile Diabetes and Work.
Brief Title: Diabetic Patients Needs in Therapeutic Education About Work. TE-DIW (Therapeutic Education of DIabetic Working People)
Acronym: ET-DIT
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL18_0824
Record Dates: First submitted 2019-03-26; First posted 2019-03-28 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Interviews — An interview will be realized with each patient in order to precise the issues they have to reconcile their diabetes and their work. Some questions will be posed to the patients and they respond as they wish.

SUMMARY:
Diabetes mellitus is an important disease around the world and the number of diabetic people increase every day. The type 1 diabetes often occurred in the youth and people have to learn to work with it and its complication. Conversely, diabetic people sometimes have trouble to manage their diabetes with working obligation. Actually, French therapeutic education don't teach how to reconcile diabetes and work. The study hypothesis is that type 1 diabetic people can be helped by therapeutic education in order to reconcile the management of their diabetes and their work. This study is a qualitative study. Interviews will help to find the needs of the type 1 diabetic patients to reconcile diabetes and work.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years old
* To be diagnosed with type 1 diabetes according to the criteria of the French High Authority of Health and confirmed by an endocrinologist
* To have paid employment with an employment contract during the study
* to be informed and having no opposition to the study

Exclusion Criteria:

* self-employed person
* to be unemployed
* To be diagnosed with an other disease wich could damage cognition or motricity and could interfere with work (cancer, neurodegenerative disorder, etc)
* To have legal guardian.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult person with a type 1 diabetes and having paid employment
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2019-04-26 (Actual); Primary Completion 2019-12-03 (Actual); Study Completion 2019-12-03 (Actual)

PRIMARY OUTCOMES:
Collection of the needs of type 1 diabetic patients in therapeutic education in order to reconcile diabetes and work. | Expected duration of interviews is around 1 hour, when no new idea appear in an interview.
  It is a qualitative study consisting of type 1 diabetic patients semi-structured interviews in order to identify and describe their needs in therapeutic education in order to reconcile diabetes and work.

CONTACTS AND LOCATIONS:
Locations (1):
- Médecine et santé au travail - Hôpital Cardiologique Louis Pradel - Groupement hospitalier Est, Bron, France

IPD SHARING:
Plan to Share IPD: No